CLINICAL TRIAL: NCT00054847
Title: CSP #474 - Radial Artery vs. Saphenous Vein Grafts in Coronary Artery Bypass Surgery (Radial Artery)
Brief Title: Radial Artery Versus Saphenous Vein Grafts in Coronary Artery Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 474
Record Dates: First submitted 2003-02-11; First posted 2003-02-13 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Cardiovascular Disease; Coronary Artery Disease
Keywords: CABG; cardiovascular; chronic diseases; clinical trial; heart; multi-site trial; prospective
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saphenous Vein Graft (Active Comparator): Saphenous Vein Graft
  Interventions: Procedure: saphenous vein graft
- Radial Artery Graft (Active Comparator): Radial Artery Graft
  Interventions: Procedure: radial artery graft

INTERVENTIONS:
Procedure: saphenous vein graft — Saphenous vein harvested from the arm is used as a conduit for CABG.
  Arms: Saphenous Vein Graft
Procedure: radial artery graft — Radial artery harvested from the arm is used as a conduit for CABG.
  Arms: Radial Artery Graft

SUMMARY:
VA patients with coronary artery disease and who have agreed to undergo coronary artery bypass graft surgery would be randomized to receive either radial artery or saphenous vein to the study vessel. The primary outcome variable is graft patency at one year.

DETAILED DESCRIPTION:
Primary Hypothesis:

Radial artery grafts will have a higher graft patency rate at one year after coronary artery bypass graft surgery (CABG) compared to saphenous vein grafts.

Secondary Hypotheses:

Determine if there are any differences in clinical outcomes, cost and quality of life in patients receiving radial artery versus saphenous vein grafts.

Intervention: 1) Saphenous vein graft. This is the standard conduit for coronary artery bypass grafting to all areas of the heart except the left anterior descending (LAD) artery. 2) Radial artery. This is the experimental conduit. Preference should be given to harvesting from the non-dominant arm.

Primary Outcomes: 1-year post CABG surgery patency rates

Study Abstract:

Although the radial artery was introduced as a potential conduit for coronary artery bypass grafting in the 1970s, enthusiasm for its use was limited by the technical difficulty of harvesting the vessel and problems with perioperative vascular spasm. In spite of this, some surgeons persisted based on their belief that arterial conduits would be better than vein grafts, in terms of long-term patency. With the development of new harvesting techniques and the introduction of calcium channel blockers to prevent vasospasm, the use of the radial artery graft has increased in recent years. This use of the radial artery as a conduit is not based on any long-term prospective data regarding its patency. However, because the VA has been a leader in defining the long-term efficacy/patency of saphenous vein and internal mammary grafts, it is appropriate for the VA to investigate radial artery grafts. In fact, the VA under its Cooperative Studies Program, is probably the only health care delivery system that has the ability to undertake this study.

Study Design:

The study is a prospective, randomized, unblinded clinical trial. The population consists of VA patients with coronary artery disease documented by coronary arteriography and who have agreed to undergo coronary artery bypass surgery. Medical conditions which could affect blood flow through the patient's arm are the main exclusion criteria. These include Raynaud's symptoms, positive Allen test, neurologic or musculoskeletal disease affecting the arm and patients with one arm.

Patients who are eligible and agree to participate in the study will be randomly assigned to receive one radial artery graft or one saphenous vein graft to the following vessels: left anterior descending if internal mammary not used, circumflex, diagonal, and right coronary artery. The surgeon will determine the subject vessel preoperatively by selecting the vessel that is suitable for grafting.

The stratification factors will be the participating hospital and which vessel is to be bypassed, left anterior descending versus all other vessels.

History, physical examination, laboratory tests, and cardiac catheterization will be performed at baseline and at one year. Follow-up clinic visits will be at two weeks, three, six, and nine months post CABG. Coronary angiography will be performed one week and one year post surgery. Quality of life and hand/leg functional status will be assessed at baseline, three months, and one year. Cost measures will be captured.

Biostatistical Considerations:

For this trial, a sample size of 874 randomized patients will be required. This will provide 90% power to detect a difference in one-year patency rates of 92% for the radial artery versus 83% for the saphenous vein and an expected one-year catheter completion rate of 65%.

This is a five year study. There will be four years of patient accrual and one year of follow-up. Nine participating VA medical centers will be expected to randomize two patients per month.

ELIGIBILITY:
Inclusion Criteria:

* Patients needing coronary artery bypass grafts.

Exclusion Criteria:

* Patients who require only a single vessel bypass and in whom the internal mammary artery will be used for that graft
* Patients with previous stripping and ligation of saphenous veins and in whom no venous conduit is available for bypass
* Patients with Raynaud's symptoms
* Patients who have a creatinine above 2.0 mg/dL or require hemodialysis
* Patients with a positive Allen test
* Patients with cardiogenic shock
* Patients who are unable to give consent
* Patients allergic to contrast material
* Patients undergoing repeat CABG or any form of robotic surgery
* Patients who do not have full use of both arms
* Patients who are pregnant
* Patients with neurologic or musculoskeletal disease affecting the arm
* Patients who refuse to participate
* Patient requires any concomitant valve operation in the mitral, aortic, or pulmonary position. Isolated tricuspid annuloplasty is acceptable, but tricuspid valve replacement excludes the patient from consideration.
* Patient requires concomitant Dor or Maze procedure
* Patient is in another research study
* No suitable radial target (there is no non-LAD vessel with a >70% stenosis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 733 (Actual)
Dates: Start 2003-02; Primary Completion 2009-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Goldman, MD, Study Chair — Southern Arizona VA Health Care System
Locations (11):
- United States (11):
  - VA Medical Center, Birmingham, Birmingham, Alabama
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock, No. Little Rock, Arkansas
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - Southeast Veterans Healthcare System, New Orleans, New Orleans, Louisiana
  - VA Boston Healthcare System, Brockton Campus, Brockton, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - New Mexico VA Health Care System, Albuquerque, Albuquerque, New Mexico
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia

REFERENCES:
- [Result] Mudumbai SC, Wagner T, Mahajan S, King R, Heidenreich PA, Hlatky M, Wallace A, Mariano ER. Vascular surgery patients prescribed preoperative beta-blockers experienced a decrease in the maximal heart rate observed during induction of general anesthesia. J Cardiothorac Vasc Anesth. 2012 Jun;26(3):414-9. doi: 10.1053/j.jvca.2011.09.027. Epub 2011 Dec 3. PMID 22138312
- [Result] Sinnott PL, Siroka AM, Shane AC, Trafton JA, Wagner TH. Identifying neck and back pain in administrative data: defining the right cohort. Spine (Phila Pa 1976). 2012 May 1;37(10):860-74. doi: 10.1097/BRS.0b013e3182376508. PMID 22127268
- [Result] Yoon J, Scott JY, Phibbs CS, Wagner TH. Recent trends in Veterans Affairs chronic condition spending. Popul Health Manag. 2011 Dec;14(6):293-8. doi: 10.1089/pop.2010.0079. Epub 2011 Nov 1. PMID 22044350
- [Result] McKellar J, Wagner T, Harris A, Oehlert M, Buckley S, Moos R. One-year outcomes of telephone case monitoring for patients with substance use disorder. Addict Behav. 2012 Oct;37(10):1069-74. doi: 10.1016/j.addbeh.2012.03.009. Epub 2012 Mar 13. PMID 22651986
- [Result] Bakaeen FG, Sethi G, Wagner TH, Kelly R, Lee K, Upadhyay A, Thai H, Juneman E, Goldman S, Holman WL. Coronary artery bypass graft patency: residents versus attending surgeons. Ann Thorac Surg. 2012 Aug;94(2):482-8; discussion 488. doi: 10.1016/j.athoracsur.2012.04.039. Epub 2012 Jun 13. PMID 22698772
- [Result] Goldman S, Sethi GK, Holman W, Thai H, McFalls E, Ward HB, Kelly RF, Rhenman B, Tobler GH, Bakaeen FG, Huh J, Soltero E, Moursi M, Haime M, Crittenden M, Kasirajan V, Ratliff M, Pett S, Irimpen A, Gunnar W, Thomas D, Fremes S, Moritz T, Reda D, Harrison L, Wagner TH, Wang Y, Planting L, Miller M, Rodriguez Y, Juneman E, Morrison D, Pierce MK, Kreamer S, Shih MC, Lee K. Radial artery grafts vs saphenous vein grafts in coronary artery bypass surgery: a randomized trial. JAMA. 2011 Jan 12;305(2):167-74. doi: 10.1001/jama.2010.1976. PMID 21224458
- [Result] Wagner TH, Holman W, Lee K, Sethi G, Ananth L, Thai H, Goldman S. The generalizability of participants in Veterans Affairs Cooperative Studies Program 474, a multi-site randomized cardiac bypass surgery trial. Contemp Clin Trials. 2011 Mar;32(2):260-6. doi: 10.1016/j.cct.2010.11.008. Epub 2010 Nov 13. PMID 21078416
- [Result] Humphreys K, Wagner TH, Gage M. If substance use disorder treatment more than offsets its costs, why don't more medical centers want to provide it? A budget impact analysis in the Veterans Health Administration. J Subst Abuse Treat. 2011 Oct;41(3):243-51. doi: 10.1016/j.jsat.2011.04.006. Epub 2011 Jun 12. PMID 21664790
- [Result] Wagner TH, Sethi G, Holman W, Lee K, Bakaeen FG, Upadhyay A, McFalls E, Tobler HG, Kelly RF, Crittenden MD, Thai H, Goldman S. Costs and quality of life associated with radial artery and saphenous vein cardiac bypass surgery: results from a Veterans Affairs multisite trial. Am J Surg. 2011 Nov;202(5):532-5. doi: 10.1016/j.amjsurg.2011.06.011. Epub 2011 Aug 26. PMID 21872209
- [Derived] Goldman S, McCarren M, Sethi GK, Holman W, Bakaeen FG, Wagner TH, Wang Y, Shih MC, Edson R; CSP #474 Investigators. Long-Term Mortality Follow-Up of Radial Artery Versus Saphenous Vein in Coronary Artery Bypass Grafting: A Multicenter, Randomized Trial. Circulation. 2022 Oct 25;146(17):1323-1325. doi: 10.1161/CIRCULATIONAHA.122.062343. Epub 2022 Oct 24. No abstract available. PMID 36279414

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicenter, randomized controlled trial conducted from February 2003 to February 2009 at 11 Veterans Affairs medical centers among 757 participants (99% men) undergoing first-time elective coronary artery bypass graft surgery.
Pre-assignment Details: The left internal mammary artery was used to preferentially graft the left anterior descending coronary artery whenever possible; the best remaining recipient vessel was randomized to radial artery vs saphenous vein graft.
Groups:
- Saphenous Vein Graft: Saphenous Vein Graft
  saphenous vein graft : Saphenous vein harvested from the arm is used as a conduit for CABG.
- Radial Artery Graft: Radial Artery Graft
  radial artery graft : Radial artery harvested from the arm is used as a conduit for CABG.
Period: Overall Study
Arm/Group | Saphenous Vein Graft | Radial Artery Graft
Started | 367 | 366
Completed | 269 | 266
Not Completed | 98 | 100

BASELINE CHARACTERISTICS:
Groups:
- Radial Artery Graft: Radial Artery
  radial artery graft : Radial artery harvested from the arm is used as a conduit for CABG.
- Total: Total of all reporting groups
Arm/Group | Saphenous Vein Graft | Radial Artery Graft | Total
Number analyzed (Participants) | 367 | 366 | 733
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8) | 61 (8) | 61.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 362 | 365 | 727
Race/Ethnicity, Customized [Number; unit: participants] — Race classification was based on prespecified categories and obtained from the patient. One patient did not specify race.
  participants
    White | 329 | 331 | 660
    Black or African American | 30 | 31 | 61
    Other | 7 | 4 | 11
    Did not specify | 1 | 0 | 1
Canadian Functional Class [Number; unit: participants] — Represents increasing angina from minimal (I) to severe incapacitating angina (IV).
  participants
    I | 75 | 79 | 154
    II | 115 | 115 | 230
    III | 132 | 127 | 259
    IV | 44 | 44 | 88
    Missing | 1 | 1 | 2
Target Vessel [Number; unit: participants]
  Left Anterior Descending | 53 | 51 | 104
  Circumflex | 215 | 203 | 418
  Right Coronary Artery | 99 | 112 | 211
Comorbidities [Number; unit: participants] — Participants may have more than one comorbidity.
  participants
    Diabetes mellitus | 153 | 154 | 307
    Hypertension | 287 | 289 | 576
    Heart Failure | 15 | 28 | 43
Previous Myocardial Infarction [Number; unit: participants] — Represents the number of patients who had a previous myocardial infarction.
  participants
    Previous Myocardial Infarction | 143 | 146 | 289
    No Previous Myocardial Infarction | 224 | 220 | 444
Smoking History [Number; unit: participants]
  Never smoked | 49 | 59 | 108
  Ex-smoker | 217 | 220 | 437
  Current smoker | 99 | 86 | 185
  Missing data | 2 | 1 | 3
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Total cholesterol level was missing for 26 patients in the saphenous vein (SV) group and 12 patients in the radial artery (RA) group.
  mg/dL | 177.2 (41.4) | 178.8 (46.8) | 177.7 (44.2)
HDL [Mean (Standard Deviation); unit: mg/dL] — HDL level was missing for 34 SV patients and 19 RA patients.
  mg/dL | 39.3 (12.2) | 38.5 (10.2) | 38.9 (11.2)
LDL [Mean (Standard Deviation); unit: mg/dL] — LDL level missing for 43 SV and 31 RA patients
  mg/dL | 105.6 (39.6) | 104.2 (38.4) | 104.9 (39.0)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] — Triglycerides level missing for 33 SV and 18 RA patients.
  mg/dL | 186.4 (118.4) | 193.0 (143.6) | 189.7 (131.8)

OUTCOME MEASURES:

1. Primary Outcome: To Compare 1-year Angiographic Patency of Radial Artery Grafts Versus Saphenous Vein Grafts in Patients Undergoing Elective Coronary Artery Bypass Graft (CABG) Surgery.
Description: The primary end point was angiographic graft patency at 1 year after coronary artery bypass surgery, defined as any opacification of distal target by injection of the graft. The window for the 1-year angiogram was 2 to 24 months. This window was chosen to capture early clinically indicated angiograms and late selective angiograms in patients who did not have symptoms. Study grafts that were occluded at 1 week after coronary artery bypass graft surgery were considered occluded at 1 year. One-year graft patency data were missing if patients whose study grafts were patent at 1 week did not undergo an angiogram within the time window or if the central angiography laboratory was not able to determine graft patency.
Time Frame: 1 year
Population: All analyses were performed according to intention to treat. The study was designed to have 90%power to detect 1-year patency rates of 92% in radial artery vs 83% in saphenous vein grafts, with a 2-sided type I error of 5% and an expected 1-year catheterization completion rate of 65%. .
Measure: Number; unit: grafts
Units Other Than Participants: Coronary Artery Bypass Grafts
Arm/Group | Saphenous Vein Graft | Radial Artery Graft
Number analyzed (Participants) | 269 | 266
Number analyzed (Coronary Artery Bypass Grafts) | 269 | 266
grafts | 269 | 266
Statistical Analysis 1: Comparison: Saphenous Vein Graft vs Radial Artery Graft; The study was designed to have 90% power to detect 1-year patency rates of 92% in radial artery vs 83% in saphenous vein grafts, with a 2-sided type I error of 5%and an expected 1-year catheterization completion rate of 65%; Test type: Superiority or Other; p = .82, Chi-squared — Multiple logistic regression analysis was used to adjust for stratification factors and characteristics that were potentially predictive of graft patency. We also performed prespecified subgroup analyses and assessed treatment subgroup interaction; We performed as-treated and per-protocol analyses & multiple imputations as sensitivity analyses to the intent-to-treat analysis on primary end point; Odds Ratio (OR) = 1.07, 95% CI 2-sided [.62 to 1.84]

2. Secondary Outcome: Death
Time Frame: Within 1 year of surgery.
Measure: Number; unit: participants
Groups:
- Radial Artery Grafts: Radial Artery Grafts
  radial artery graft: Radial artery harvested from the arm is used as a conduit for CABG.
Arm/Group | Saphenous Vein Graft | Radial Artery Grafts
Number analyzed (Participants) | 367 | 366
participants | 7 | 9
Statistical Analysis 1: Comparison: Saphenous Vein Graft vs Radial Artery Grafts; Test type: Superiority or Other; p = .61, Chi-squared

3. Secondary Outcome: Myocardial Infarction
Time Frame: Within 1 year of bypass surgery
Measure: Number; unit: participants
Groups:
- Arm 1: Saphenous Vein Graft
  saphenous vein graft: Saphenous vein harvested from the arm is used as a conduit for CABG.
- Arm 2: Radial Artery
  radial artery graft: Radial artery harvested from the arm is used as a conduit for CABG.
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 367 | 366
participants | 5 | 4
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p > .99, Chi-squared

4. Secondary Outcome: Stroke
Time Frame: Within 1 year of bypass surgery
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 367 | 366
participants | 6 | 7

ADVERSE EVENTS:
Time Frame: From time of consent through follow-up.
Description: The verbatim description was used to classify events by Body System affected (System Organ Class or SOC) and to group using a common medical term (Preferred Term or PT).
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 172/367 | 158/366
Other Adverse Events (participants affected / at risk) | 152/367 | 161/366
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=367) | Arm 2 (N=366)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 2 (2) | 2 (2)
Angiogram (Investigations) | 2 (2) | 0 (0)
Angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic bypass (Surgical and medical procedures) | 3 (4) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Arterial repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Aspiration pleural cavity (Investigations) | 0 (0) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 11 (11) | 14 (20)
Atrial flutter (Cardiac disorders) | 2 (2) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Blood culture positive (Investigations) | 1 (1) | 1 (1)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 7 (7) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 6 (10) | 9 (14)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 4 (5) | 4 (4)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 2 (2) | 1 (1)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (2) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Catheterisation cardiac (Investigations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 4 (4)
Cellulitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 6 (7) | 3 (3)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 19 (20) | 17 (18)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Claustrophobia (Psychiatric disorders) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 2 (2)
Coagulation time prolonged (Investigations) | 1 (1) | 0 (0)
Colectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colonoscopy (Investigations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 3 (3) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 2 (3)
Coronary artery occlusion (Cardiac disorders) | 3 (3) | 3 (3)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cyst (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 2 (2)
Debridement (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Dermatitis infected (Infections and infestations) | 0 (0) | 1 (1)
Detoxification (Surgical and medical procedures) | 1 (1) | 0 (0)
Device damage (General disorders) | 1 (1) | 0 (0)
Device function test (Investigations) | 2 (2) | 1 (1)
Device occlusion (General disorders) | 0 (0) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Drug rehabilitation (Surgical and medical procedures) | 0 (0) | 1 (1)
Drug screen positive (Investigations) | 1 (1) | 0 (0)
Drug therapy changed (Surgical and medical procedures) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Endarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Gastric dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hernia (General disorders) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Implant site pain (General disorders) | 0 (0) | 1 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 2 (2) | 4 (5)
Incision site cellulitis (Infections and infestations) | 5 (5) | 2 (2)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incisional drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Laryngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leg amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Living in residential institution (Social circumstances) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Mechanical ventilation (Surgical and medical procedures) | 2 (2) | 3 (3)
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0)
Medical device complication (General disorders) | 1 (1) | 0 (0)
Medical observation (Investigations) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 5 (6)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 2 (2)
Neurological decompensation (Nervous system disorders) | 0 (0) | 1 (1)
Neurological symptom (Nervous system disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Parotid gland inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Penile prosthesis insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 5 (5) | 4 (4)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
Peripheral artery angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Peripheral artery bypass (Surgical and medical procedures) | 3 (3) | 3 (3)
Peripheral artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 2 (2)
Peripheral revascularisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 2 (2) | 3 (3)
Plastic surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 16 (16)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 4 (4)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Post procedural complication (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Post procedural drainage (Surgical and medical procedures) | 1 (2) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (5) | 3 (3)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Post procedural stroke (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative thoracic procedure compli (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 14 (16) | 12 (14)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Psychiatric evaluation (Investigations) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 3 (3)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Self-injurious ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Splenectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Stent placement (Surgical and medical procedures) | 1 (1) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis in device (General disorders) | 1 (1) | 0 (0)
Toe amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Transplant evaluation (Investigations) | 1 (1) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Typical aura without headache (Nervous system disorders) | 1 (1) | 0 (0)
Unevaluable event (General disorders) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 4 (4) | 3 (4)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound drainage (Surgical and medical procedures) | 3 (3) | 0 (0)
Wound infection (Infections and infestations) | 1 (2) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=367) | Arm 2 (N=366)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal wall mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 4 (4) | 2 (2)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 6 (6)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 3 (5)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Angiopathy (Vascular disorders) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Anxiety postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Arthrectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 16 (16) | 15 (16)
Atrial flutter (Cardiac disorders) | 3 (3) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 9 (9)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 4 (4)
Biopsy kidney (Investigations) | 0 (0) | 1 (1)
Biopsy liver (Investigations) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 4 (4) | 4 (4)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 1 (2) | 0 (0)
Brachial plexus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 4 (4)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breath sounds abnormal (Investigations) | 0 (0) | 1 (1)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Bunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Cardiac enzymes increased (Investigations) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac stress test (Investigations) | 1 (1) | 0 (0)
Cardiac stress test normal (Investigations) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 2 (2)
Cataract (Eye disorders) | 1 (1) | 2 (2)
Catheter removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 5 (6)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 4 (4) | 0 (0)
Chest pain (General disorders) | 9 (13) | 13 (17)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Coagulation time prolonged (Investigations) | 1 (1) | 0 (0)
Coccidioidomycosis (Infections and infestations) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Crepitations (General disorders) | 0 (0) | 1 (1)
Cystoscopy (Investigations) | 1 (1) | 0 (0)
Debridement (Surgical and medical procedures) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 5 (5) | 7 (7)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Device breakage (General disorders) | 1 (1) | 1 (1)
Device function test (Investigations) | 1 (1) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Dizziness exertional (Nervous system disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (7)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Ear injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Echocardiogram (Investigations) | 1 (1) | 1 (1)
Effusion (General disorders) | 0 (0) | 1 (1)
Elective procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Electrocardiogram ST segment elevation (Investigations) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Entropion (Eye disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Exposure to chemical pollution (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 2 (2)
Eye allergy (Eye disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 6 (7)
Fatigue (General disorders) | 0 (0) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Groin infection (Infections and infestations) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Haematocrit decreased (Investigations) | 2 (3) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 3 (3)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (11) | 10 (13)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 (7) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 11 (13) | 9 (10)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 9 (9) | 17 (19)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 5 (5) | 4 (4)
Hypothyroidism (Endocrine disorders) | 3 (3) | 4 (4)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (6)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Implantable defibrillator insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Incision site abscess (Infections and infestations) | 1 (1) | 2 (2)
Incision site cellulitis (Infections and infestations) | 3 (3) | 11 (12)
Incision site complication (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Incision site erythema (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Incision site infection (Infections and infestations) | 2 (2) | 1 (1)
Incision site oedema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Incisional drainage (Surgical and medical procedures) | 2 (2) | 2 (2)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Influenza immunisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Infusion site phlebitis (General disorders) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Injection site infection (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 4 (4)
Insulin resistance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 4 (4) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Joint arthroplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Joint injection (Surgical and medical procedures) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Keloid scar (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Local swelling (General disorders) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Macular oedema (Eye disorders) | 1 (1) | 0 (0)
Medical device complication (General disorders) | 3 (3) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Mononeuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Nerve root compression (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 2 (2)
Onychomycosis (Infections and infestations) | 2 (2) | 4 (4)
Ophthalmological examination (Investigations) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 1 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 3 (3)
Pain (General disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (3) | 2 (2)
Patient restraint (Surgical and medical procedures) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Peripheral nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Physical assault (Social circumstances) | 1 (1) | 0 (0)
Physical examination (Investigations) | 3 (3) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 13 (14)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Postoperative thoracic procedure complica (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 11 (12) | 12 (12)
Presyncope (Nervous system disorders) | 1 (1) | 2 (2)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Puncture site haemorrhage (General disorders) | 1 (1) | 1 (1)
Purulent discharge (Infections and infestations) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 5 (5) | 2 (2)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 3 (3)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (2)
Renal mass (Renal and urinary disorders) | 1 (1) | 1 (1)
Respiratory depth decreased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 2 (4)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (2) | 2 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Scar pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Somnambulism (Psychiatric disorders) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Suture removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Suture rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Swelling (General disorders) | 1 (1) | 1 (2)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Systolic hypertension (Vascular disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tenderness (General disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombophlebitis (Vascular disorders) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tinea infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Transfusion (Surgical and medical procedures) | 1 (2) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ulcer (General disorders) | 0 (0) | 1 (1)
Unevaluable event (General disorders) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 7 (7)
Urethral stenosis (Renal and urinary disorders) | 2 (4) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 6 (6) | 5 (5)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Urological examination (Investigations) | 0 (0) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 2 (2) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 3 (3)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Vital signs measurement (Investigations) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Wound infection pseudomonas (Infections and infestations) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
There was more disease in the radial artery grafts at 1 week and at 1 year. There is more spasm or string sign in radial artery grafts. Study was conducted predominantly in men. Data show lower vein graft patency when endoscopic harvesting was used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes